CLINICAL TRIAL: NCT02461589
Title: Dose-finding of Semaglutide Administered Subcutaneously Once Daily Versus Placebo and Liraglutide in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-4191; 2014-003196-39 (EudraCT Number); U1111-1159-4923 (Other: WHO)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (13):
- Semaglutide 0.05 mg/day (Experimental)
  Interventions: Drug: semaglutide
- Liraglutide 0.3 mg/day (Active Comparator)
  Interventions: Drug: liraglutide
- Placebo 50 µL (Placebo Comparator)
  Interventions: Drug: placebo
- Semaglutide 0.05/0.1 mg/day (Experimental)
  Interventions: Drug: semaglutide
- Liraglutide 0.3/0.6 mg/day (Active Comparator)
  Interventions: Drug: liraglutide
- Placebo 50/100 µL (Placebo Comparator)
  Interventions: Drug: placebo
- Semaglutide 0.05/0.1/0.2 mg/day (Experimental)
  Interventions: Drug: semaglutide
- Liraglutide 0.3/0.6/1.2 mg/day (Active Comparator)
  Interventions: Drug: liraglutide
- Placebo 50/100/200 µL (Placebo Comparator)
  Interventions: Drug: placebo
- Semaglutide 0.05/0.1/0.2/0.3 mg/day (Experimental)
  Interventions: Drug: semaglutide
- Liraglutide 0.3/0.6/1.2/1.8 mg/day (Active Comparator)
  Interventions: Drug: liraglutide
- Placebo 50/100/200/300 µL (Placebo Comparator)
  Interventions: Drug: placebo
- Semaglutide flexible escalation from 0.05 mg/day to 0.3 mg/day (Experimental)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Administered subcutaneously ( s.c., under the skin) once daily. All subjects will follow a 4-week dose-escalation regimen except subjects who received semaglutide flexible dosing.
  Arms: Semaglutide 0.05 mg/day; Semaglutide 0.05/0.1 mg/day; Semaglutide 0.05/0.1/0.2 mg/day; Semaglutide 0.05/0.1/0.2/0.3 mg/day; Semaglutide flexible escalation from 0.05 mg/day to 0.3 mg/day
Drug: liraglutide — Administered subcutaneously ( s.c., under the skin) once daily. All subjects will follow a 4-week dose-escalation regimen.
  Arms: Liraglutide 0.3 mg/day; Liraglutide 0.3/0.6 mg/day; Liraglutide 0.3/0.6/1.2 mg/day; Liraglutide 0.3/0.6/1.2/1.8 mg/day
Drug: placebo — Administered subcutaneously ( s.c., under the skin) once daily.
  Arms: Placebo 50 µL; Placebo 50/100 µL; Placebo 50/100/200 µL; Placebo 50/100/200/300 µL

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate dose-finding of semaglutide administered subcutaneously once daily versus placebo and liraglutide in subjects with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 18 years at the time of signing informed consent.
* Subjects should be on stable diabetes treatment consisting of diet and exercise with or without metformin (at least 1500 mg daily or maximum tolerated dose documented in the patient medical record) for at least 90 days prior to screening
* HbA1c (glycosylated haemoglobin): 53-86 mmol/mol (7.0-10.0%) (both inclusive)
* BMI: 25.0 - 40.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Simultaneous participation in any other clinical trial of an investigational medicinal product
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods throughout the trial including the 7 weeks follow-up period (adequate contraceptive measures as required by local regulation or practice). Germany: Only highly effective methods of birth control are accepted (i.e. one that results in less than 1% per year failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine device), or sexual abstinence or vasectomised partner. United Kingdom: Adequate contraceptive measures are defined as established use of oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device or intrauterine system, barrier methods of contraception (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository), female sterilisation, male sterilisation (where partner is sole partner of subject), or true abstinence (when in line with preferred and usual lifestyle)
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before screening (an exception is short-term insulin treatment for acute illnesses for a total of below or equal to 14 days)
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days or on an frequent basis) known to affect weight or glucose metabolism (e.g. orlistat, thyroid hormones, corticosteroids)
* History of pancreatitis (acute or chronic)
* Screening calcitonin above or equal to 50 ng/L
* Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN2) or Medullary Thyroid Carcinoma (MTC)
* Severe to moderate renal impairment defined as GFR, estimated below 60 ml/min/1.73 m^2 as per CKD-EPI (Chronic Kidney Disease Epidemiology)
* Within the past 180 days before screening any of the following: Myocardial infarction, stroke or hospitalisation for unstable angina and/or transient ischemic attack
* Currently planned coronary, carotid or peripheral artery revascularisation
* Patients presently classified as being in New York Heart Association (NYHA) Class III or IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2016-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (136):
- United States (74):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Coronado, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Riverside, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Van Nuys, California
  - Novo Nordisk Investigational Site, Vista, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Hartford, Connecticut
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Ponte Vedra, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Evanston, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Newton, Kansas
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Marrero, Louisiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Belzoni, Mississippi
  - Novo Nordisk Investigational Site, Bridgeton, Missouri
  - Novo Nordisk Investigational Site, Kalispell, Montana
  - Novo Nordisk Investigational Site, Elkhorn, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Hopewell Junction, New York
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Delaware, Ohio
  - Novo Nordisk Investigational Site, Dublin, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Corvallis, Oregon
  - Novo Nordisk Investigational Site, Downingtown, Pennsylvania
  - Novo Nordisk Investigational Site, Media, Pennsylvania
  - Novo Nordisk Investigational Site, Smithfield, Pennsylvania
  - Novo Nordisk Investigational Site, Uniontown, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Hodges, South Carolina
  - Novo Nordisk Investigational Site, Mt. Pleasant, South Carolina
  - Novo Nordisk Investigational Site, Old Point Station, South Carolina
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Johnson City, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Carrollton, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Missouri City, Texas
  - Novo Nordisk Investigational Site, New Braunfels, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Waco, Texas
  - Novo Nordisk Investigational Site, Bountiful, Utah
  - Novo Nordisk Investigational Site, Clinton, Utah
  - Novo Nordisk Investigational Site, Riverton, Utah
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Saint Stefan
  - Novo Nordisk Investigational Site, Vienna
- Canada (7):
  - Novo Nordisk Investigational Site, Coquitlam, British Columbia
  - Novo Nordisk Investigational Site, Moncton, New Brunswick
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
  - Novo Nordisk Investigational Site, Strathroy, Ontario
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Pointe-Claire, Quebec
- Czechia (8):
  - Novo Nordisk Investigational Site, Benešov
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Liberec
  - Novo Nordisk Investigational Site, Náchod
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Police nad Metují
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Trutnov
- Germany (9):
  - Novo Nordisk Investigational Site, Eisenach
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Sulzbach-Rosenberg
- Malaysia (5):
  - Novo Nordisk Investigational Site, George Town
  - Novo Nordisk Investigational Site, Klang, Selangor
  - Novo Nordisk Investigational Site, Kota Bharu
  - Novo Nordisk Investigational Site, Seremban
  - Novo Nordisk Investigational Site, Seri Manjung
- Russia (7):
  - Novo Nordisk Investigational Site, Dzerzhinskiy
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Smolensk
  - Novo Nordisk Investigational Site, Syktyvkar
  - Novo Nordisk Investigational Site, Voronezh
- Serbia (5):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
  - Novo Nordisk Investigational Site, Zaječar
- South Africa (5):
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Midrand, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Middleburg, Mpumalanga
- United Kingdom (13):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Bexhill-on-Sea
  - Novo Nordisk Investigational Site, Blackburn
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Chesterfield, Derbyshire
  - Novo Nordisk Investigational Site, Devon
  - Novo Nordisk Investigational Site, Harrogate, North Yorkshire
  - Novo Nordisk Investigational Site, Hinckley
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Sidcup
  - Novo Nordisk Investigational Site, Truro

REFERENCES:
- [Result] Lingvay I, Desouza CV, Lalic KS, Rose L, Hansen T, Zacho J, Pieber TR. A 26-Week Randomized Controlled Trial of Semaglutide Once Daily Versus Liraglutide and Placebo in Patients With Type 2 Diabetes Suboptimally Controlled on Diet and Exercise With or Without Metformin. Diabetes Care. 2018 Sep;41(9):1926-1937. doi: 10.2337/dc17-2381. Epub 2018 Jul 19. PMID 30026333
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 139 sites in 10 countries as follows:
  Austria: 3 sites; Canada: 8 sites; Czech Republic: 9 sites; Germany:
  7 sites; Malaysia: 5 sites; Russian Federation: 7 sites; Serbia: 9 sites; South Africa: 7 sites; United Kingdom: 13 sites; United States: 71 sites.
Pre-assignment Details: Of the 706 subjects randomised in the trial, 705 were exposed to trial products and 1 randomised subject withdrew prior to exposure.
Groups:
- Semaglutide 0.05 mg/Day: Participants received semaglutide 0.05 mg subcutaneous (sc) injection once daily for 26 weeks. Semaglutide injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals.
- Semaglutide 0.1 mg/Day: Participants received semaglutide 0.05 mg sc injection once daily for 4 weeks followed by semaglutide 0.1 mg once daily upto week 26. Semaglutide injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals.
- Semaglutide 0.2 mg/Day: Participants received semaglutide 0.05 mg sc injection once daily for 4 weeks followed by semaglutide 0.1 mg once daily for next 4 weeks and then semaglutide 0.2 mg once daily upto week 26. Semaglutide injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals.
- Semaglutide 0.3 mg/Day: Participants received semaglutide 0.05 mg sc injection once daily for 4 weeks followed by semaglutide 0.1 mg once daily for next 4 weeks followed by 0.2 mg once daily for next 4 weeks and then semaglutide 0.3 mg once daily upto week 26. Semaglutide injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals.
- Liraglutide 0.3 mg/Day: Participants received liraglutide 0.3 mg sc injection once daily for 26 weeks. Liraglutide injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals.
- Liraglutide 0.6 mg/Day: Participants received liraglutide 0.3 mg sc injection once daily for 4 weeks followed by liraglutide 0.6 mg once daily upto week 26. Liraglutide injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals.
- Liraglutide 1.2 mg/Day: Participants received liraglutide 0.3 mg sc injection once daily for 4 weeks followed by liraglutide 0.6 mg once daily for next 4 weeks and then liraglutide 1.2 mg once daily upto week 26. Liraglutide injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals.
- Liraglutide 1.8 mg/Day: Participants received liraglutide 0.3 mg sc injection once daily for 4 weeks followed by liraglutide 0.6 mg once daily for next 4 weeks followed by liraglutide 1.2 mg once daily for next 4 weeks and then liraglutide 1.8 mg once daily upto week 26. Liraglutide injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals.
- Placebo: Participants received placebo (the volume matched the volume used for the specific dose of semaglutide or liraglutide) sc injection once daily upto 26 weeks. Placebo injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals.
- Semaglutide Flexible: Participants received semaglutide 0.05 mg sc injection once daily for 4 weeks followed by semaglutide 0.1 mg once daily for next 4 weeks followed by 0.2 mg once daily for next 4 weeks and then semaglutide 0.3 mg once daily upto week 26. Semaglutide injection was administered in the thigh, abdomen, or upper arm, preferably around the same time of the day irrespective of meals. Participants were allowed to follow a more flexible dose-escalation regimen based on gastrointestinal tolerability. Semaglutide dose levels could be reduced in participants with poor gastrointestinal tolerability depending on investigator's assessment.
Period: Overall Study
Arm/Group | Semaglutide 0.05 mg/Day | Semaglutide 0.1 mg/Day | Semaglutide 0.2 mg/Day | Semaglutide 0.3 mg/Day | Liraglutide 0.3 mg/Day | Liraglutide 0.6 mg/Day | Liraglutide 1.2 mg/Day | Liraglutide 1.8 mg/Day | Placebo | Semaglutide Flexible
Started | 64 | 63 | 65 | 63 | 64 | 64 | 64 | 65 | 129 | 65
Exposed | 64 | 63 | 65 | 63 | 64 | 64 | 64 | 65 | 129 | 64
Completed | 58 | 61 | 60 | 58 | 62 | 61 | 58 | 60 | 123 | 60
Not Completed | 6 | 2 | 5 | 5 | 2 | 3 | 6 | 5 | 6 | 5
Not completed — Withdrawal by Subject | 5 | 1 | 3 | 2 | 1 | 2 | 1 | 3 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 3 | 1 | 1 | 3 | 1 | 3 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Unclassified | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Missing follow-up information | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal from trial before exposure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the full analysis set (FAS) which included all randomised subjects who had received at least 1 dose of either semaglutide, liraglutide or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.05 mg/Day | Semaglutide 0.1 mg/Day | Semaglutide 0.2 mg/Day | Semaglutide 0.3 mg/Day | Liraglutide 0.3 mg/Day | Liraglutide 0.6 mg/Day | Liraglutide 1.2 mg/Day | Liraglutide 1.8 mg/Day | Placebo | Semaglutide Flexible | Total
Number analyzed (Participants) | 64 | 63 | 65 | 63 | 64 | 64 | 64 | 65 | 129 | 64 | 705
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.53 (9.8) | 57.51 (10.0) | 58.37 (9.58) | 54.76 (9.66) | 57.20 (10.78) | 59.45 (9.77) | 53.73 (11.35) | 55.82 (9.19) | 57.08 (9.25) | 54.81 (9.70) | 56.67 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 22 | 31 | 35 | 32 | 30 | 32 | 57 | 28 | 326
  Male | 33 | 35 | 43 | 32 | 29 | 32 | 34 | 33 | 72 | 36 | 379
HbA1c (glycosylated haemoglobin) [Mean (Standard Deviation); unit: percentage of HbA1c] | 7.87 (0.71) | 7.91 (0.83) | 7.96 (0.82) | 8.23 (0.80) | 8.06 (0.86) | 8.12 (0.81) | 8.14 (0.87) | 8.07 (0.85) | 8.12 (0.87) | 8.10 (0.91) | 8.06 (0.84)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 9.26 (2.60) | 8.97 (2.22) | 9.20 (2.28) | 9.67 (2.56) | 9.32 (2.54) | 9.34 (2.33) | 9.91 (2.70) | 9.18 (2.45) | 9.67 (2.98) | 9.82 (2.66) | 9.45 (2.59)
Body weight [Mean (Standard Deviation); unit: kg] | 93.44 (18.27) | 92.40 (17.20) | 98.07 (17.92) | 94.82 (17.84) | 92.25 (17.48) | 92.68 (16.46) | 96.67 (18.28) | 93.40 (19.34) | 93.98 (17.75) | 95.29 (15.43) | 94.28 (17.61)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 133.70 (15.14) | 130.97 (14.92) | 131.34 (12.55) | 132.08 (11.69) | 134.02 (11.30) | 132.41 (12.37) | 134.20 (12.73) | 131.02 (11.86) | 132.17 (14.26) | 132.70 (12.74) | 132.43 (13.10)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 80.06 (8.90) | 79.71 (8.56) | 80.48 (8.87) | 81.41 (8.05) | 81.83 (6.98) | 81.28 (6.90) | 82.98 (6.94) | 80.66 (7.62) | 80.98 (8.00) | 81.89 (8.40) | 81.11 (7.96)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Estimated mean change from baseline in HbA1c at week 26. The data were analysed for the "on-treatment until rescue medication" observation period which includes observations recorded at or after date of first dose of trial product and not after the last dose of trial product plus the 7-day visit window or date of initiation of rescue therapy.
Time Frame: Week 0, week 26
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Semaglutide 0.05 mg/Day | Semaglutide 0.1 mg/Day | Semaglutide 0.2 mg/Day | Semaglutide 0.3 mg/Day | Liraglutide 0.3 mg/Day | Liraglutide 0.6 mg/Day | Liraglutide 1.2 mg/Day | Liraglutide 1.8 mg/Day | Placebo | Semaglutide Flexible
Number analyzed (Participants) | 64 | 63 | 65 | 63 | 64 | 64 | 64 | 65 | 129 | 64
percentage of glycosylated haemoglobin | -0.97 (0.85) | -1.30 (1.03) | -1.65 (0.79) | -1.96 (0.95) | -0.50 (0.93) | -0.88 (0.90) | -0.86 (0.92) | -1.32 (0.78) | -0.05 (0.90) | -1.72 (0.97)
Statistical Analysis 1: Comparison: Semaglutide 0.05 mg/Day vs Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.04, 95% CI 2-sided [-1.30 to -0.77]
Statistical Analysis 2: Comparison: Semaglutide 0.1 mg/Day vs Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.34, 95% CI 2-sided [-1.61 to -1.08]
Statistical Analysis 3: Comparison: Semaglutide 0.2 mg/Day vs Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.69, 95% CI 2-sided [-1.95 to -1.42]
Statistical Analysis 4: Comparison: Semaglutide 0.3 mg/Day vs Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.86, 95% CI 2-sided [-2.12 to -1.60]

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Estimated mean change from baseline in FPG at week 26. The data were analysed for the "on-treatment until rescue medication" observation period which includes observations recorded at or after date of first dose of trial product and not after the last dose of trial product plus the 7-day visit window or date of initiation of rescue therapy.
Time Frame: Week 0, Week 26
Population: Full analyses set. For "Semaglutide flexible arm", data was available only for 63 subjects.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 0.05 mg/Day | Semaglutide 0.1 mg/Day | Semaglutide 0.2 mg/Day | Semaglutide 0.3 mg/Day | Liraglutide 0.3 mg/Day | Liraglutide 0.6 mg/Day | Liraglutide 1.2 mg/Day | Liraglutide 1.8 mg/Day | Placebo | Semaglutide Flexible
Number analyzed (Participants) | 64 | 63 | 65 | 63 | 64 | 64 | 64 | 65 | 129 | 63
mmol/L | -2.09 (1.96) | -2.08 (2.23) | -2.64 (2.07) | -3.53 (2.20) | -1.33 (2.06) | -1.56 (1.74) | -1.51 (2.41) | -1.92 (2.34) | -0.54 (2.45) | -3.40 (2.84)

3. Secondary Outcome: Body Weight Change
Description: The data were analysed for the "on-treatment until rescue medication" observation period which includes observations recorded at or after date of first dose of trial product and not after the last dose of trial product plus the 7-day visit window or date of initiation of rescue therapy.
Time Frame: Week 0, Week 26
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Semaglutide 0.05 mg/Day | Semaglutide 0.1 mg/Day | Semaglutide 0.2 mg/Day | Semaglutide 0.3 mg/Day | Liraglutide 0.3 mg/Day | Liraglutide 0.6 mg/Day | Liraglutide 1.2 mg/Day | Liraglutide 1.8 mg/Day | Placebo | Semaglutide Flexible
Number analyzed (Participants) | 64 | 63 | 65 | 63 | 64 | 64 | 64 | 65 | 129 | 64
kg | -2.75 (2.82) | -4.36 (4.24) | -6.70 (4.57) | -8.23 (5.34) | -1.48 (3.06) | -1.81 (3.06) | -1.78 (3.41) | -3.68 (4.26) | -1.22 (3.42) | -6.60 (4.98)

4. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: as for outcome 3
Time Frame: Week 0, Week 26
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 0.05 mg/Day | Semaglutide 0.1 mg/Day | Semaglutide 0.2 mg/Day | Semaglutide 0.3 mg/Day | Liraglutide 0.3 mg/Day | Liraglutide 0.6 mg/Day | Liraglutide 1.2 mg/Day | Liraglutide 1.8 mg/Day | Placebo | Semaglutide Flexible
Number analyzed (Participants) | 64 | 63 | 65 | 63 | 64 | 64 | 64 | 65 | 129 | 64
mmHg
  Systolicblood pressure | -5.74 (12.30) | -2.77 (13.21) | -4.25 (12.24) | -9.85 (11.58) | -3.77 (9.79) | -3.20 (10.89) | -4.69 (12.73) | -2.99 (11.94) | -2.34 (11.40) | -6.62 (14.02)
  Diastolic blood pressure | -0.60 (8.78) | 0.66 (8.26) | -1.62 (9.38) | -4.02 (8.56) | -1.77 (7.37) | -1.89 (8.20) | -0.60 (6.78) | 0.63 (8.13) | -0.61 (8.50) | -1.69 (8.25)

ADVERSE EVENTS:
Time Frame: From baseline up to week 33.
Description: Safety analysis set (SAS) included all randomised subjects exposed to at least one dose of trial product. Subjects in the SAS would contribute to the evaluation "as treated". Treatment-emergent adverse events (TEAEs) were defined as events recorded from the first dose of trial product and until completion of the post-treatment follow-up visit (7 weeks).
Arm/Group | Semaglutide 0.05 mg/Day | Semaglutide 0.1 mg/Day | Semaglutide 0.2 mg/Day | Semaglutide 0.3 mg/Day | Liraglutide 0.3 mg/Day | Liraglutide 0.6 mg/Day | Liraglutide 1.2 mg/Day | Liraglutide 1.8 mg/Day | Placebo | Semaglutide Flexible
Serious Adverse Events (participants affected / at risk) | 7/64 | 3/63 | 2/65 | 2/63 | 1/64 | 2/64 | 2/64 | 7/65 | 0/129 | 4/64
Other Adverse Events (participants affected / at risk) | 31/64 | 34/63 | 39/65 | 42/63 | 33/64 | 27/64 | 35/64 | 35/65 | 0/129 | 44/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.05 mg/Day (N=64) | Semaglutide 0.1 mg/Day (N=63) | Semaglutide 0.2 mg/Day (N=65) | Semaglutide 0.3 mg/Day (N=63) | Liraglutide 0.3 mg/Day (N=64) | Liraglutide 0.6 mg/Day (N=64) | Liraglutide 1.2 mg/Day (N=64) | Liraglutide 1.8 mg/Day (N=65) | Placebo (N=129) | Semaglutide Flexible (N=64)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular graft (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.05 mg/Day (N=64) | Semaglutide 0.1 mg/Day (N=63) | Semaglutide 0.2 mg/Day (N=65) | Semaglutide 0.3 mg/Day (N=63) | Liraglutide 0.3 mg/Day (N=64) | Liraglutide 0.6 mg/Day (N=64) | Liraglutide 1.2 mg/Day (N=64) | Liraglutide 1.8 mg/Day (N=65) | Placebo (N=129) | Semaglutide Flexible (N=64)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 3 (4) | 1 (1) | 2 (3) | 1 (1) | 3 (5) | 2 (2) | 4 (13) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 2 (4) | 3 (7) | 5 (6) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 4 (7)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (5) | 4 (4) | 1 (2) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 2 (2) | 2 (4) | 3 (3) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 4 (5)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (11) | 5 (7) | 0 (0) | 3 (3) | 1 (2) | 7 (7) | 0 (0) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 4 (5) | 3 (3) | 1 (2) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 7 (7) | 6 (6) | 8 (8) | 2 (3) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 7 (10) | 10 (13) | 10 (15) | 16 (29) | 5 (5) | 5 (9) | 5 (8) | 8 (16) | 0 (0) | 11 (22)
Dizziness (Nervous system disorders) | 2 (4) | 4 (6) | 2 (2) | 3 (4) | 0 (0) | 3 (4) | 1 (1) | 4 (5) | 0 (0) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 1 (6) | 5 (7) | 5 (8) | 6 (6) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Fatigue (General disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (5) | 4 (6) | 1 (1) | 0 (0) | 2 (3) | 2 (3) | 1 (2) | 0 (0) | 6 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (8) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Headache (Nervous system disorders) | 7 (17) | 8 (30) | 4 (13) | 7 (11) | 5 (7) | 3 (11) | 10 (16) | 4 (8) | 0 (0) | 7 (14)
Hypertension (Vascular disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 3 (4) | 3 (5) | 4 (5) | 7 (7) | 0 (0) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (12) | 6 (7) | 4 (4) | 5 (6) | 4 (5) | 3 (3) | 5 (7) | 5 (6) | 0 (0) | 10 (11)
Nausea (Gastrointestinal disorders) | 11 (16) | 12 (20) | 14 (22) | 16 (22) | 6 (7) | 7 (11) | 7 (11) | 13 (18) | 0 (0) | 25 (35)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 3 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 2 (2) | 1 (1) | 7 (7) | 6 (6) | 1 (1) | 2 (3) | 5 (6) | 0 (0) | 4 (6)
Vomiting (Gastrointestinal disorders) | 6 (10) | 4 (13) | 6 (9) | 6 (8) | 1 (1) | 7 (10) | 1 (1) | 5 (8) | 0 (0) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property